CLINICAL TRIAL: NCT04137315
Title: Project Aura: Data Collection for a Home Monitoring Solution for Patients With Anaemia to Evaluate Delivery of Treatment
Brief Title: Project Aura: Home Trial of a Home-based Monitoring Service
Status: Completed | Type: Observational
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IRAS: 272300
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Blood measurement — Single fingerprick to measure haemoglobin and haematocrit measurements using a potential haemoglobin home monitoring system.

SUMMARY:
This is a data collection study to compare diagnostic methods of a prototype of a home monitoring device against laboratory testing in the hospital.

DETAILED DESCRIPTION:
The device/monitoring system being developed measures the haemoglobin and haematocrit levels in blood from a single drop of blood. By measuring these blood parameters, participants are able to monitor their haemoglobin level at home.

The use of the device will take place in the participant's home to simulate what the investigators believe will be the ideal location for people who would prefer to self-manage their condition.

This study is a data collection study to evaluate the performance of the prototype.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age.
* Adequate english to participate in training sessions and use the analyser.
* Patients of the study site who are currently undergoing treatment for anaemia of CKD with ESAs.
* Patients who are not pregnant.
* Patients who do not have a bleeding disorder.
* Patients willing to perform self-tests 2-3 times a week.
* Patients capable of providing informed consent before attending training.
* Patients or patients with a carer capable of fine manipulation of the device and its consumables.
* Patients or patients with a carer who own a smartphone which can download the app related to this study.
* Patients or patients with carers who do not have eyesight limitations to be able to read the instructions on the screen of the prototype device.
* Patients who are not expected to have to start dialysis treatment during the course of this study.

Exclusion Criteria:

* Does not have adequate English to participate in training or use the analyser without an interpreter.
* Patients of the study site who are not currently undergoing anaemia treatment with ESAs.
* Patients of the study site not willing to perform self-tests 2-3 times a week.
* Patients of the study site not capable of providing consent or have a suitable, legally acceptable representative present to provide consent before the trial.
* Patients who are pregnant.
* Patients with a bleeding disorder.
* Patients or their nominated carers who are not capable of fine manipulation of the device and its consumables.
* Neither patients or their nominated carers do not own a smartphone which can install the app related to this study.
* Patients or their nominated carers with eyesight limitations to not be able to read the instructions on the screen of the prototype device.
* Patients who are expected to start dialysis treatment during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from the study site.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Quantitative capture of measurement system | 6 months
  Data collection for evaluation of measurement system

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Bhandari, FHEA, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Hull University Teaching Hospitals NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Study data will be pseudonymous (shared with the research & clinical team). Participant data is only seen by the research nurse for contacting, updating and travel reimbursement purposes.